CLINICAL TRIAL: NCT04954690
Title: Structured Program of Exercise for Recipients of Kidney Transplantation
Acronym: SPaRKT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-28357
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Kidney Transplant; Complications; Dialysis; Complications; Physical Disability; Frailty Syndrome
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: This is an exercise intervention. Therefore participation and coaching cannot be masked. In order to ensure safety, the primary nephrologist and dialysis clinic will be informed of patients participation in the trial. However, they will not be involved with coaching or assessing outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Placebo Comparator): Patients randomized to usual care will receive recommendations for exercise based on the Surgeon General's recommendations for physical activity among adults as well as the American Heart Association and American College of Sports Medicine recommendations for older individuals or individuals with chronic conditions. These guidelines are applicable to this patient population. Patients will not receive coaching but will receive accelerometers to obtain data for comparison to the intervention groups at each time point (baseline, 8 weeks, and 3 months post-KT).
  Interventions: Behavioral: Usual Care
- Weekly Coaching (Active Comparator): Weekly coaching per the SPaRKT protocol with titrated increases in physical activity and resistance exercise
  Interventions: Behavioral: Structured Program of exercise for Recipients of Kidney Transplantation (WC)
- Weekly Coaching + Caregiver Participation (Active Comparator): Weekly coaching per the SPaRKT protocol with titrated increases in physical activity and resistance exercise with the addition of caregiver participation to promote adherence and engagement
  Interventions: Behavioral: Structured Program of exercise for Recipients of Kidney Transplantation (WC + CG)

INTERVENTIONS:
Behavioral: Structured Program of exercise for Recipients of Kidney Transplantation (WC) — Structured Program of exercise for Recipients of Kidney Transplantation (weekly coaching)
  Other Names: WC
  Arms: Weekly Coaching
Behavioral: Structured Program of exercise for Recipients of Kidney Transplantation (WC + CG) — Structured Program of exercise for Recipients of Kidney Transplantation (weekly coaching + caregiver participation)
  Other Names: WC+CG
  Arms: Weekly Coaching + Caregiver Participation
Behavioral: Usual Care — Usual Care
  Arms: Usual Care

SUMMARY:
Older patients with end- stage kidney disease (ESKD) are at very high risk for functional impairment. Kidney transplantation (KT) has the potential to ameliorate the detrimental effects of ESKD on physical activity and functional status. However, KT alone may not meet the full extent of this potential, particularly for older or more impaired adults. In fact, activity declines immediately post-KT and fails to return to expected levels even 5 years post-KT. Older patients waitlisted for KT (most of whom are on dialysis) are therefore reliant on their pre-KT levels of exercise, which are also predictive of post-KT mortality.

"Prehabilitation" has been used in other surgical populations to minimize functional loss, and a structured exercise program may be beneficial in the pre- KT setting. However, few waitlisted patients are able to participate in typical exercise interventions due to barriers such as severe fatigue. Older patients have additional barriers such as further mobility impairment and requiring substantial caregiver support. Therefore for older living donor kidney transplant candidates, it is necessary to address issues such as specifics of coaching, timing, and importantly, incorporate caregiver participation.

The overall objective of this proposal is to adapt a previously developed 8- week, home- based, structured exercise program among older (≥50 years) dialysis patients awaiting living donor KT, with a focus on caregiver involvement. The investigators will trial the exercise program as compared to usual care. The investigators will then pilot the refined intervention in a total of 72 patient-caregiver dyads, 48 of whom will undergo the proposed intervention (24 with caregiver participation, 24 without). The primary outcomes for the pilot will be change in physical performance and activity from baseline to after the intervention, along with measurements of exploratory quality of life outcomes. In addition, the investigators will measure these same outcomes at 3- months post KT to evaluate for a durable effect of the intervention. An additional post-transplantation outcome of interest will be number of days hospitalized within 3 months of transplantation.

DETAILED DESCRIPTION:
The investigators will conduct a randomized clinical trial of 72 eligible participants to test SPaRKT versus usual care. The primary outcome will be ascertained at completion of the 8-week program and at 3 months post-KT. This study will provide the successful completion rate of weekly coaching as well as estimates of the impact of SPaRKT as compared to usual care. This proposal is powered primarily for change in physical function and change in walking as determined by accelerometers.

Prior to the trial, the investigators will first conduct an "adaptation" phase where study personnel recruit 10-15 paired patient-caregiver dyads to work out any logistical issues with the intervention and work on incorporating caregiver participation. This initial adaptation phase will involve focus groups of each individual wave. In addition, participants and caregivers in the adaptation portion of the study will be asked to give weekly feedback on the intervention, delivered through semi-scripted qualitative interviews of participants and caregivers. Among the items the investigators will attempt to ascertain will be: appropriate length of discussion, preferred method (phone vs video), and preferred feedback during health coaching. The investigators will conduct a final focus group interview of all participants in the adaptation phase to provide consensus on SPaRKT prior to the randomized controlled trial.

Pre-intervention: At time of enrollment, study personnel will provide information to all patients and caregivers on: 1) potential benefits of exercise and increasing activity, 2) the association between poor physical function and adverse outcomes in ESKD and specifically in KT, 3) the typical course of changes in physical function and activity post-KT, 4) general recommendations for activity. The investigators will review patient records for dialysis prescription, laboratory results, comorbid conditions, and medications. All participants will be given a Fitbit Inspire 2 (Fitbit, Inc.) accelerometer and instructed in calibration and use. The Fitbit Inspire 2 is similar to the older model (now discontinued) Fitbit Zip, in that it can be placed on a lower extremity. The Fitbit Zip has been validated in older, community-dwelling adults, and is accurate in individuals with slower walking. Participants will be asked to record activity for a one week lead-in period immediately prior to baseline assessment.

SPaRKT (intervention): Participants and caregivers will be guided through video exercises adapted for hemodialysis and peritoneal dialysis patients from the Strong for Life™ series of exercise videos to determine starting resistance band level, demonstrate proper positioning, and provide instruction on adjusting resistance. Each participant will engage in the videos a second time to enforce proper positioning. The Strong for Life™ videos were developed for sedentary older adults with physical disability. The adapted video series will consist of 11 exercises incorporating movement patterns used in daily activities. Some of these exercises use resistance bands. Study personnel will provide Thera-bands™ in 3 levels of resistance to each participant. Starting resistance and subsequent progression will be adapted from the Strong for Life™ protocol; a health coach will ask participants to increase the level of resistance when they are able to perform 12-15 repetitions of an exercise without loss of proper execution. Participants will be instructed to exercise using the these exercise videos 3 times per week for the 8-week intervention period, a dose found to be safe and effective in improving functional status among older adults post-hip fracture.

A health coach will be assigned to each participant in SPaRKT as the primary contact for counseling, feedback, and assistance. The health coach will call the participant once per week using a semi-structured script which will be refined during the adaptation phase. For Aim 1 and for the WC+CG group in Aims 2 and 3, caregivers will be included on calls. Participants will be counseled to increase their average daily steps by 10% for the next week's goal, starting from their baseline activity during the lead-in period. Participants will be instructed to adhere to participation in the exercise program, including with the Strong for Life™ video. Participants in SPaRKT will have recommendations for gradual increases of exercise per their individual health coach as guided by the protocol for 8 weeks. Afterwards, they will be asked to maintain exercise until KT.

Caregiver participation: For the Weekly Coaching + Caregiver Participation (WC+CG) arm in the intervention, caregivers will be asked to participate along with the older adult they are paired with. For the first week, personnel will request that caregivers keep track of patient activity logs and participate in weekly coaching sessions. During these sessions, a health coach will ask caregivers to plan how their patient can reach next week's activity and exercise goals. For later weeks, a health coach will encourage caregivers to 1) perform mid-week checks to ensure that patients will meet their targets, 2) take and increase number of walks with the patient in a stepwise fashion and 3) accompany the patient for exercise sessions.

Participant randomization. For the trial, participants will be randomized to SPaRKT (weekly coaching, WC: N=24, weekly coaching + caregivers, WC+CG: N=24) or usual care (N=24) with more patients in SPaRKT in order to have more experience working through the logistics of the intervention. Random assignments will be generated prior to the study using a computerized randomization scheme with assignments placed into sequentially numbered sealed envelopes. Assignment will be performed after living donor KT is scheduled and baseline assessment of outcomes has been performed.

For the WC+CG group, caregivers in the WC+CG group will be given guidelines based on feedback from the adaptation phase.

Usual Care: Patients randomized to usual care will receive recommendations for exercise based on the Surgeon General's recommendations for physical activity among adults5 as well as the American Heart Association and American College of Sports Medicine recommendations for older individuals or individuals with chronic conditions. These guidelines are applicable to this patient population. Patients will not receive coaching but will receive accelerometers to obtain data for comparison to the intervention groups at each time point (baseline, 8 weeks, and 3 months post-KT).

ELIGIBILITY:
Inclusion Criteria:

* On hemodialysis or peritoneal dialysis
* Age ≥ 50 years
* SPPB score ≤ 10
* Telephone access
* Internet access
* Having a living donor kidney

Exclusion Criteria:

* Already in an exercise program
* Non-English speakers

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) | baseline, 8 weeks (post-program completion), approximately 20 weeks (3-months post-KT)
  The Short Physical Performance Battery (SPPB) is a composite score ranging from 0-12, with three tests which measure: 1) gait speed, 2) timed sit to stand, and 3) balance. Each individual component can be scored from 0-4 with a total score of 0-12, with higher numbers representing better physical performance.
Change in Step Count | baseline, 8 weeks (post-program completion), approximately 20 weeks (3-months post-KT)
  Change in Step Count (determined by accelerometer). Step counts will be measured as continuous variables, with higher step count meaning a higher level of activity.

SECONDARY OUTCOMES:
Change in 6 minute walk distance (6MWD) | baseline, 8 weeks (post-program completion), approximately 20 weeks (3-months post-KT)
  The six-minute walk test (6MWT) measures the distance in meters an individual is able to walk over a total of six minutes on a hard, flat surface. Higher distances achieved are considered better.
Change in Grip Strength | baseline, 8 weeks (post-program completion), approximately 20 weeks (3-months post-KT)
  Grip strength will be measured by handheld dynamometer (kg force), with increased kg of force representing greater grip strength.
Change in Short Form-36 (SF-36) score | baseline, 8 weeks (post-program completion), approximately 20 weeks (3-months post-KT)
  The Short Form-36 (SF-36) is a generic health score to measure global functioning consisting of 36 questions measuring eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. The scores are transformed to a range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health.
Change in Center for Epidemiological Studies- Depression (CES-D) score | baseline, 8 weeks (post-program completion), approximately 20 weeks (3-months post-KT)
  The Center for Epidemiological Studies- Depression (CES-D) is a 20-item measure that asks caregivers to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Change in Dialysis Symptoms Index (DSI) score | baseline, 8 weeks (post-program completion), approximately 20 weeks (3-months post-KT)
  The Dialysis Symptoms Index (DSI) contains 30 items, each of which targets a specific physical or emotional symptom. Patients are asked to report the presence (yes/no) of each symptom at any time during the previous 7 days. Using a five-point Likert scale (1 = "not at all bothersome" to 5 = "bothers very much"), the severity of each symptom reported as being present is assessed by asking patients to rate the degree to which the symptom is bothersome. Scores can therefore range from 0 to 150, with higher scores being representative of more symptoms and more bothersome symptoms.
Change in lower urinary tract symptoms (LUTS questionnaire) | baseline, 8 weeks (post-program completion), approximately 20 weeks (3-months post-KT)
  This questionnaire measures lower urinary tract symptoms of interest, including urinary frequency, incontinence, hesitance, and bother, with higher scores indicating more or more bothersome symptoms.
Change in Montreal Cognitive Assessment (MoCA) | baseline, 8 weeks (post-program completion), approximately 20 weeks (3-months post-KT)
  Change in cognition per the Montreal Cognitive Assessment (MoCA). The MoCA is a is a brief 30-question test that takes around 10 to 12 minutes to complete and helps assess people for dementia. Scores range from 0 to 30 with scores of 26 and above are generally considered "normal" with scores below 26 implying some degree of cognitive impairment.
Days hospitalized after transplantation | approximately 20 weeks (3-months post-KT)
  Days hospitalized after transplantation (within 90 days). Inpatient days specifically will be measured.
Days in rehabilitation after transplantation | approximately 20 weeks (3-months post-KT)
  Days in rehabilitation after transplantation (within 90 days). Days in skilled nursing facility or rehabilitation centers specifically will be measured. Outpatient rehabilitation or physical therapy will be considered separately.

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Sheshadri, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- Connie Frank Center for Kidney Transplantation at the University of California, San Francisco Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications after deidentification will be shared (texts, tables, figures, appendices, etc).
Supporting Information: Study Protocol
Time Frame: Beginning 6 months after publication and ending 36 months after publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose, for individual participant data meta-analyses.